CLINICAL TRIAL: NCT04981808
Title: The Diabetes teleMonitoring of Patients in Insulin Therapy (DiaMonT) Trial: Study Protocol for a Randomized Controlled Trial
Brief Title: Diabetes teleMonitoring of Patients in Insulin Therapy
Acronym: DiaMonT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Steno Diabetes Center Sjaelland (Other Government); Novo Nordisk A/S (Industry); Glooko (Industry); DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Peter Vestergaard, MD, professor, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-20200068
Record Dates: First submitted 2021-06-08; First posted 2021-07-29 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Type 2 Diabetes Treated With Insulin
Keywords: Diabetes; Insulin; Telemedicine; Telehealth; Telemonitoring; CGM; Adherence
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemonitoring (Experimental): The subjects will be telemonitored. All subject will use a CGM, a fit bit, and a smart pen during the entire trial period. Staff at the endocinology clinics will monitor the data and contact the subjects continuously throughout the trial (depending on the individual needs of each subject)
  Interventions: Device: Telemonitoring
- Usual Care (No Intervention): The subjects will wear a blinded CGM the first and final 20 days of the trial. The subjects will use a blinded smart pen throughout the trial period. Hence, the subjects are unable to see their measured data during the trial, and they will not be monitored.

INTERVENTIONS:
Device: Telemonitoring — Telemonitoring of CGM and insulin pen data
  Arms: Telemonitoring

SUMMARY:
The trial is an open-label randomized controlled trial. Patients with T2D on insulin therapy will be randomized to a telemonitoring group (intervention) and a usual care group (control). The telemonitoring group will use various devices at home. Hospital staff will monitor their data for a period of three months.

DETAILED DESCRIPTION:
The DiaMonT trial is an open-label randomized controlled trial with a trial period of three months conducted. The trial will be conducted in two sites in Denmark: Steno Diabetes Center North Jutland and Steno Diabetes Center Zealand. Patients with T2D on insulin therapy will be randomized (1:1) to a telemonitoring group (intervention) or a usual care group (control). The telemonitoring group will use an insulin pen, an activity tracker, a CGM, and a smartphone application throughout the trial period. Hospital staff (lab technicians and nurses) will monitor the telemonitoring groups' data and contact the subjects by telephone repeatedly throughout the trial period. The usual care group will use a blinded CGM the first and last 20 days of the trial and will use a blinded insulin pen for the entire period. The usual care groups' data will not be monitored during the trial.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* T2D diagnosis for ≥ 12 months
* Residence in Region North Denmark or Region Zealand
* In treatment with insulin
* Being able to use a smartphone along with the other devices to be used in the trial
* Able to understand and read Danish.

Exclusion Criteria:

* Pregnancy or breastfeeding,
* Major surgery planned during the trial period
* Participation in other trials
* Terms that, in the opinion of the investigator or subinvestigators, render the participant unfit to conduct the trial, including lack of understanding of the trial or lack of physical or cognitive ability to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
CGM time in range | At baseline to three months after randomization
  Change in CGM time in range (3,9-10,0 mmol/L)

SECONDARY OUTCOMES:
Concentration of HbA1c | At baseline to three months after randomization
  Change in HbA1c
Total daily units of insulin | At baseline to three months after randomization
  Change in total daily dose of insulin (units)
Time below CGM range | At baseline to three months after randomization
  Change in time below range (CGM)
Time above CGM range | At baseline to three months after randomization
  Change in time above range (CGM)

OTHER OUTCOMES:
Number of CGM days worn | During the intervention
  Number of days that the subjects wear the CGM
CGM percentage of time active | During the intervention
  Percentage of time that the CGM is active
Mean glucose | At baseline to three months after randomization
  Mean glucose levels (mmol/l) measured by CGM
Glycemic variability | At baseline to three months after randomization
  Glycemic variability - percentage of cofficient of variation
Time in hyperglycemia | At baseline to three months after randomization
  Time in hyperglycemia (>13,9 mmol/L)
Time in hypoglycemia | At baseline to three months after randomization
  Time in hypoglycemia (<3,0 mmol/L)
Episodes of hyperglycemia | At baseline to three months after randomization
  Number of episodes of hyperglycemia (>13,9 mmol/L)
Episodes of hypoglycemia | At baseline to three months after randomization
  Number of episodes in hypoglycemia
Use of the telemonitoring equipment | Through study completion, an average of 3 months
  The frequency of use of the telemonitoring equipment
Telemonitoring usability | Immediately after the intervention
  Telemonitoring satisfaction and usability measured by the Telemonitoring Usability Questionnaire (TUQ). Minimum value =1, maximum value =7. A higher score = a better outcome
Diabetes-related quality of life | From baseline to three months after randomization
  Diabetes-related quality of life measured by the DIDP Questionnaire. Ranges from "very negative" to "very positive"
Health-related quality of life | From baseline to three months after randomization
  Health-related quality of life measured by the Short Form 12 (SF-12). Options are not numeric

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hangaard S, Kronborg T, Hejlesen O, Aradottir TB, Kaas A, Bengtsson H, Vestergaard P, Jensen MH. The Diabetes teleMonitoring of patients in insulin Therapy (DiaMonT) trial: study protocol for a randomized controlled trial. Trials. 2022 Dec 7;23(1):985. doi: 10.1186/s13063-022-06921-6. PMID 36476605